CLINICAL TRIAL: NCT05040633
Title: Evaluating the Clinical Effectiveness of Adjunct Low-level Laser Therapy (ECEALT) in the Management of Chronic Low-Back Pain: A Long-Term, Double-Blind, Randomized Control Trial in Physiotherapy Clinics in Ontario, Canada
Brief Title: The ECEALT Chronic Low Back Pain Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Health Rehab and Research Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V2/0518
Record Dates: First submitted 2021-07-10; First posted 2021-09-10 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Chronic Low-back Pain
Keywords: Laser Therapy; Low Back Pain; Randomized Control Trial
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to three groups and provided with one of the following interventions: (i) Low Level Laser Therapy (LLLT) therapy in combination with standard exercise therapy (Arm 1), (ii) sham LLLT therapy in combination with standard exercise therapy (Arm 2), or (iii) exercise therapy alone (Arm 3).
  Participants will receive treatment three times per week for four consecutive weeks (i.e., each participant will receive a total of 12 treatment sessions; see section 2, Trial Design).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization codes will be generated by a member of the trial team who is not involved in the day-to-day running of the trial, nor will they be involved in future data analysis. Each participant's randomized code will be kept in a sealed envelope to be opened only by the assessor during the first trial visit. The assessor and patients will be blinded to treatment allocation but physiotherapists offering treatment will not be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Level Laser Therapy + standard exercise therapy (Experimental): This group of participants will first receive the standard therapy of strengthening and stretching exercises followed by the Low Lever Laser Therapy.
  Interventions: Device: BTL 4110 Smart Laser Therapy Equipment (BTL Industries Ltd, United Kingdom (UK)); Other: Standard Exercise Therapy
- Sham Low Level Laser Therapy + standard exercise therapy (Sham Comparator): This group of participants will first receive the standard therapy of strengthening and stretching exercises followed by a sham Low Level Laser Therapy (LLLT). The laser equipment will be deactivated and not switched on.
  Interventions: Device: BTL 4110 Smart Laser Therapy Equipment (BTL Industries Ltd, United Kingdom (UK)); Other: Standard Exercise Therapy
- Standard Exercise Therapy (Active Comparator): Trial participants in this group will only receive the standard exercise therapy. The exercise therapy will consist of strengthening and stretching exercises.
  Interventions: Other: Standard Exercise Therapy

INTERVENTIONS:
Device: BTL 4110 Smart Laser Therapy Equipment (BTL Industries Ltd, United Kingdom (UK)) — Participants will receive 12 LLLT sessions during the course of the trial, thrice weekly for 4 consecutive weeks. Doses will be as per the recommendations of the Wold Association of Laser Therapy.
  Arms: Low Level Laser Therapy + standard exercise therapy; Sham Low Level Laser Therapy + standard exercise therapy
Other: Standard Exercise Therapy — Exercise therapy will consist of strengthening and stretching exercises. At each visit, participants will perform each of the exercises under the supervision of a licensed physiotherapist.

SUMMARY:
The primary objective of this double-blind randomized control trial (RCT) is to evaluate the clinical effectiveness of LLLT as adjunctive therapy to standard exercise treatment in patients with non-specific chronic LBP. Specifically, the study will aim to evaluate the effectiveness of adjunct LLLT in the reduction of pain in patients as well as determine its long-term functional outcomes.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most common musculoskeletal disorders and the leading cause of years lived with disability worldwide with significant socioeconomic impacts. Around 10-15 % of LBP patients develop chronic symptoms lasting more than 3 months, and this is considered chronic, with the causes often being "non-specific" with no identifiable causes. Despite the availability of medication-based protocols, the management of non-specific chronic LBP (NSCLBP) is an increasing challenge to clinicians and their patients. Adjunctive therapy can play an important role in the treatment of NSCLBP. In recent decades, low-level laser therapy (LLLT) has been widely used to relieve pain caused by different musculoskeletal disorders. Though widely used and reported as a safe, non-invasive treatment with minimal side effects; reported therapeutic outcomes of LLLT are varied and conflicting, due in part to methodological concerns, lack of data and unclear results.

ELIGIBILITY:
Inclusion Criteria:

* are 18-65 years with the ability to give informed consent
* report with non - specific chronic low back pain, which is defined as pain of >3 months duration that occurs in the lumbosacral area of the spine, which may or not have the characteristics of limiting the patient's range of movements, and is not attributable to a recognizable, known pathology (e.g., infection, tumor, osteoporosis, lumbar spine fracture, structural deformity, inflammatory disorder, radicular syndrome, or cauda equina syndrome).
* are experiencing pain measured using the Quadruple Visual Analogue Scale between 4 and 7 at the time of assessment will be included to keep homogeneity of pain.

Exclusion Criteria:

* are under 18 years, and those over 65 years of age
* have had past fractures of the bone structures of the spine
* have had previous surgery of the spine
* have a history of previous surgery of the spine or vertebra; spondylosis, spinal stenosis, lumbar disc herniation
* use pacemakers (cardiac or brain)
* are pregnant, or those who plan to become pregnant during the course of the study
* have acute and/or chronic cardiovascular diseases
* have dermatological conditions in the area of irradiation and/or inflammatory skin lesions
* have tattoo/tattoos around the area of irradiation
* have any sensory deficits as defined by the World Health Organization's working definition
* are sensitive/allergic to phototherapy
* have neurological disorders as defined by the World Health Organization's working definition
* are taking anti-inflammatories or analgesic or psychotropic medications
* have any current infections
* have a history of drug abuse, either recreational, over the counter or prescription over the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain using the Quadruple Visual Analog Scale | Weeks 1, 2, 3, 6, 8, 12, 26 and 52
  The change in Pain measured using the Quadruple Visual Analog Scale (QVAS) measured at weeks 1, 2, 3, 6, 8, 12, 26 and 52. Pain reduction measured on a 10-point Likert scale from 0 (no pain) to 10 (worst possible pain). Overall score interpreted based on QVAS scoring manual of <50(Low intensity) and >50 (high intensity).
Change in Pain using the McGill Pain Questionnaire | Weeks 1, 2, 3, 6, 8, 12, 26 and 52
  The change in Pain measured using the McGill Pain Questionnaire measured at weeks 1, 2, 3, 6, 8, 12, 26 and 52. Pain reduction assessed based on an overall score ranging from 0 (would not be seen in a person with true pain) to 78(seen in a person with the greatest pain).
Change in Pain using the Brief Pain Inventory | Weeks 1, 2, 3, 6, 8, 12, 26 and 52
  The change in Pain measured using the Brief Pain Inventory measured at weeks 6, 8, 12, 26 and 52. Pain reduction assessed based on an overall score ranging from 0 (no pain or does not interfere) to 10(pain as bad as be imagined or completely interferes).

SECONDARY OUTCOMES:
Reliance on medication for pain management using the Brief Pain Inventory | Weeks 1, 2, 3, 6, 8, 12, 26 and 52
  Reliance on medication for pain management measured using the Brief Pain Inventory (short form) measured at weeks 6, 8, 12, 26 and 52. Pain reduction assessed based on an overall score ranging from 0% (no relief) to 100% (complete relief).
Mean Pain Free Days/Months using the Brief Pain Inventory | Weeks 1, 2, 3, 6, 8, 12, 26 and 52
  Mean Pain Free Days measured using the Brief Pain Inventory measured at weeks 6, 8, 12, 26 and 52. Pain reduction assessed based on an overall score ranging from 0 (no pain or does not interfere) to 10(pain as bad as can be imagined or completely interferes).
Fear of Pain measured using the McGill Pain Questionnaire | Weeks 1, 2, 3, 6, 8, 12, 26 and 52
  Fear of pain measured using the McGill Pain Questionnaire at weeks 1, 2, 3, 6, 8, 12, 26 and 52. Fear of Pain assessed on a 3-point scale from 1(fearful), 2 (frightful) or 3 (terrifying).
Frequency of Low Back Pain Episodes assessed using patients personal daily pain records | Weeks 1, 2, 3, 6, 8, 12, 26 and 52
  Frequency of LBP episodes during trial measured using patients personal daily pain records at weeks 1, 2, 3, 4, 6, 8, 12, 26 and 52. Each episode of pain recorded as a single occurrence.
Mean number of days absent from work measured using patients personal daily pain record | Weeks 1, 2, 3, 6, 8, 12, 26 and 52
  Mean number of days absent from work measured using patients personal daily pain records at weeks 1, 2, 3, 4, 6, 8, 12, 26 and 52. Not being able to work completely due to pain within a work day recorded as a single day, while working for less than 4 hours due to pain recorded as partial work day.

CONTACTS AND LOCATIONS:
Overall Officials: Hammad Qazi, PhD, Principal Investigator — Health and Rehab Research Inc
Locations (1):
- Health and Rehab Research Inc., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared externally or with other researchers.